CLINICAL TRIAL: NCT01142375
Title: Development and Exploration of the Feasibility of Using Locally Synthesized Small Molecule Inhibitors to Treat Human Acute Leukemia Cells
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Hsingjin Eugene Liu, MD PhD, Taipei Medical University WanFang Hospital
Other Study IDs: Leukemia-001
Record Dates: First submitted 2010-06-09; First posted 2010-06-11 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bone Marrow
Oversight: Data Monitoring Committee: No

SUMMARY:
Acute leukemias are commonly seen in elderly and have no effective therapy. In recent years, small molecule inhibitors have shown a tremendous promise in cancer treatment such as chronic myeloid leukemia and lung cancer. Thus, in this proposal, we intend to use our novel patented "indole" compound to conjugated with hydroxamic acid in histone deacetylases inhibitor, suberoylanilide hydroxamic acid and further modify its structure to generate novel small-molecule anticancer compounds. By screening acute leukemic cell lines, we will look for compounds that have shown potential for future drug development. In our preliminary studies, we have identified a novel compound, MPT0E001, to have marked growth inhibitory activity, induce apoptosis and downregulate c-Myc protein level. We intend to use MPT0E001 as a basis to develop novel compounds and test them in multiple leukemic cell lines and primary leukemia samples (Specific aim 1) and identify the mechanisms for downregulation of c-Myc and other pathways such as NF-kappaB and Akt (Specific aim 2). Once we have identified the lead compounds, we will use murine model to assess the acute toxicity profiles in different dose ranges and examine the effects of blood counts and vital organs. After toxicity study, we will test the lead compounds using in vivo xenogenic murine model using both cell lines and primary leukemia. Using this approach, we hope to develop novel compounds that are able to be used in future leukemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Acute Myeloid Leukemia

Exclusion Criteria:

* Hematologic malignancies other than AML

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Acute Leukemia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-04

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Gjin Eugene Liu, Principal Investigator — Taipei Medical University WanFang Hospital